CLINICAL TRIAL: NCT01007604
Title: Efficacy Study of a Peristaltic Pulse Pneumatic Device in the Treatment of Claudication
Brief Title: Treatment of Claudication With a Peristaltic Pulse Pneumatic Device
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: NormaTec Industries LP (Industry)
Responsible Party: Sharon Besso, ARNP, White River Junction VAMC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21975
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Intermittent Claudication
Keywords: claudication; pneumatic compression device
MeSH Terms: conditions — Intermittent Claudication | interventions — Exercise Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and lifestyle counselling (Active Comparator): Patients will receive standard recommendations for ambulatory exercise and standard educational discussion of risk factor control, including smoking cessation.
  Interventions: Other: Exercise and lifestyle counseling
- PCD with peristaltic pulse waveform (Experimental): Daily use for two hours
  Interventions: Device: Peristaltic pulse PCD

INTERVENTIONS:
Device: Peristaltic pulse PCD — Daily use for two hours
  Other Names: NormaTec PCD; Exercise and lifestyle counselling
  Arms: PCD with peristaltic pulse waveform
Other: Exercise and lifestyle counseling — Patients will receive standard recommendations for ambulatory exercise and standard educational discussion of risk factor control, including smoking cessation.
  Other Names: Ambulatory exercise; Smoking cessation counseling
  Arms: Exercise and lifestyle counselling

SUMMARY:
The purpose of this study is to evaluate the efficacy of a non-invasive peristaltic pulse pneumatic device (PCD) in the treatment of intermittent claudication in patients having documented peripheral arterial disease (PAD). The pneumatic device to be studied is FDA approved for the treatment of venous disease. While anecdotal evidence exists supporting a decrease in claudication symptoms, there are no previously published data on studies employing this compression device in the treatment of arterial disease. The investigators' primary hypothesis is that patients randomized to the intervention arm of the trial will experience an increase in mean walking ability as compared to the group receiving medical standard of care.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a common disorder, affecting 12% of adults older than 50 years of age. Approximately one third of these patients experience intermittent claudication, defined as pain in the thigh or calf muscles during walking and that resolves with rest. Lower extremity pain is often severe enough to significantly limit ambulation, forcing many patients to seek medical care. Current treatments include two FDA-approved medications, supervised walking programs, arterial angioplasty and/or stent placement, and open arterial bypass surgery. The problem is that noninvasive treatments are oftentimes ineffective, while invasive treatments are effective but expensive.

A non-invasive lower extremity treatment that has shown success in treating lymphedema and venous insufficiency will be studied during this protocol to assess its effects on claudication symptoms. Half of the participants in this prospective, single-center randomized controlled trial will be treated with a pneumatic compression device in a home treatment program, while half will receive standard medical therapy. If effective, potential benefits are high, providing relief of personal disability and avoidance of costly surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Consistent claudication symptoms for at least 6 months
* ABIs at rest as follows: 0.5>ABI<0.8 minimally on one leg

Exclusion Criteria:

* Refuses to consent
* Unlikely to be compliant with protocol
* Unable to perform treadmill test
* Current use of Cilostazol (Pletal) or Pentoxyphylline (Trental)
* Lower extremity surgery or endovascular procedure within the last 3 months
* Currently has a non-healing wound on either leg
* DVT in the past 3 months
* Unstable hypertension, angina, uncontrolled glucose levels
* Participating in a supervised exercise regimen
* Claudication medications regime changed within the last 3 months
* Diagnosis of Raynaud's Disease
* Requires a custom fabricated boot appliance
* Single limb amputees meeting inclusion criteria may participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Peak walking time (in seconds) during a graded-protocol treadmill test | initial; 3 months; 6 months

SECONDARY OUTCOMES:
Claudication onset time (in seconds) during a graded-protocol treadmill test | initial; 3 months; six months
Walking Impairment Questionnaire, including pain subscale, speed subscale and stair climbing subscale | initial; 3 months; 6 months
Ankle-Brachial Index (ABI) | initial; 3 months; 6 months
Integumentary changes as evaluated by photographs of lower extremity hair pattern and great toenail growth | initial; 3 months; 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon R Besso, MS, ARNP, Principal Investigator — White River Junction Veterans Affairs Medical Center; Joseph P Duggan, DPM, Principal Investigator — White River Junction Veterans Affairs Medical Center
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States